CLINICAL TRIAL: NCT01906385
Title: A Dual Phase 1/2, Investigator Initiated Study to Determine the Maximum Tolerated Dose, Safety, and Efficacy of 186Rhenium Nanoliposomes (186RNL) in Recurrent Glioma (CTRC# 12-02)
Brief Title: Maximum Tolerated Dose, Safety, and Efficacy of Rhenium Nanoliposomes in Recurrent Glioma (ReSPECT)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Plus Therapeutics (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRC 12-02; 14-450X (Other: UT Health San Antonio); 20141749 (Other: WIRB); 1R01CA235800-01A1 (NIH)
Record Dates: First submitted 2012-01-11; First posted 2013-07-24 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Glioma
Keywords: Glioma; Brain Tumor; Radiotherapy; Glioblastoma; Recurrent Glioblastoma; Rhenium; Rhenium Nanoliposome; Brain Cancer; GBM; High Grade Glioma; Glioblastoma Multiform; Grade IV Astrocytoma
MeSH Terms: conditions — Glioma; Brain Neoplasms; Glioblastoma

STUDY DESIGN:
Intervention Model Description: Phase 1:
  • Single arm, prospective study utilizing a modified Fibonacci dose escalation scheme.
  Phase 2:
  • Single arm, prospective study utilizing a non-DLT dose obtained from the dose escalation portion of IND 116117, NIH-NCI Grant (22.3 mCi (total 186RNL activity) at a concentration of 2.5 mCi/mL and 8.8 mL total volume).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 186Rhenium Liposome Treatment (Experimental): Arm
  Phase I:
  Experimental: Dose Escalation for Cohorts 1-8 Each participant will receive a single administration of 186RNL. At each dose level, a minimum of three to a maximum of six participants will be enrolled.
  If no dose limiting toxicity is observed in the initial three participants, then the next higher dose level cohort will open for enrollment.
  The dose escalation scheme will follow a modified Fibonacci dose escalation scheme as shown below:
  COHORT ACTIVITY Cohort 1 (1.0 mCi) Cohort 2 (2.0 mCi) Cohort 3 (4.0 mCi) Cohort 4 (8.0 mCi) Cohort 5 (13.4 mCi) Cohort 6 (22.3 mCi) Cohort 7 (31.2 mCi) Cohort 8 (41.5 mCi)
  Phase 2:
  Single arm, prospective study utilizing a non-DLT dose obtained from the dose escalation portion of IND 116117, NIH-NCI Grant (22.3 mCi (total 186RNL activity) at a concentration of 2.5 mCi/mL and 8.8 mL total volume).
  Interventions: Drug: Rhenium Liposome Treatment

INTERVENTIONS:
Drug: Rhenium Liposome Treatment — At the time of stereotactic biopsy a catheter will be placed within the tumor using stereotactic guidance. Once the patient has adequately recovered from the procedure as determined by the neurosurgeon, 186RNL will be infused through the CED catheter at the predetermined dose. Spectroscopic imaging will then be obtained at predefined time points to visualize the distribution of the 186RNL as well as calculated the actual dose retained within the tumor. Patients will be monitored longitudinally for evidence of toxicity and response by MRI.
  Other Names: Rhenium-186 NanoLiposome

SUMMARY:
This is a multi-center, sequential cohort, open-label, volume and dose escalation study of the safety, tolerability, and distribution of 186RNL given by convection enhanced delivery to patients with recurrent or progressive malignant glioma after standard surgical, radiation, and/or chemotherapy treatment. The study uses a modified Fibonacci dose escalation, followed by an expansion at the maximum tolerated dose (MTD) to determine efficacy. The starting absorbed dose is 1mCi in a volume of 0.660mL.

DETAILED DESCRIPTION:
The Phase I portion of the clinical study evaluates a single dose of 186RNL (radionuclide clinical study drug) administered through a convection enhanced delivery catheter (CED catheter) in participants with recurrent Glioma (GBM). The clinical study treatment consists of a single administered dose of 186RNL per participant. The clinical study will include the evaluation of multiple separate dose levels (dose escalation). Three to six participants may be treated at each dose. The maximum number of participants to be enrolled in the study is approximately 21. The clinical study treatment will be administered, following CED placement, by the clinical study physician. Participants will be followed for up to 36 months after the clinical study drug is administered.

The Phase II portion of the clinical study is a multicenter, single arm, prospective study utilizing a non-DLT dose obtained from the dose escalation portion of IND 116117, NIH-NCI Grant (22.3 mCi (total 186RNL activity) at a concentration of 2.5 mCi/mL and 8.8 mL total volume). The maximum number of participants to be enrolled in the Phase II study is approximately 34. The clinical study treatment will be administered, following CED placement, by the clinical study physician. Participants will be followed for up to 36 months after the clinical study drug is administered.

The U.S. Food and Drug Administration (FDA) has not approved 186RNL for this specific disease.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee.
3. Histologically confirmed Grade III/IV recurrent Glioma (following 2021 WHO CNS5 glioma nomenclature, e.g., Astrocytoma, IDH-mutant grade 3 or 4; Glioblastoma, IDH-wildtype grade 4).
4. Progression by RANO criteria or other clinically accepted neurooncology evaluation, following standard treatment options with known survival benefit for any recurrence (e.g., surgery, temozolomide, radiation, and tumor treating fields). Patient may be included in study if medically unable or unwilling to follow standard treatment options for any recurrence.
5. Patients who receive treatment with antiepileptic medications must have a two-week history of stable dose of antiepileptic without seizures prior to study start (dosing).
6. Patients with corticosteroid requirements to control cerebral edema must be maintained at a stable or decreasing dose for a minimum of two weeks without progression of clinical symptoms prior to study start (dosing).
7. Patients with Grade III/IV Glioma (following 2021 WHO CNS5 glioma nomenclature, e.g., Astrocytoma, IDH-mutant grade 3 or 4; Glioblastoma, IDH-wildtype grade 4) which falls within the treatment field volume.
8. ECOG performance status of 0 to 2; Karnofsky Performance Status ≥ 60.
9. Life expectancy of at least 2 months.
10. Acceptable liver function:

    1. Bilirubin ≤ 1.5 times upper limit of normal
    2. AST (SGOT) and ALT (SGPT) ≤ 3.0 times upper limit of normal (ULN)
11. Acceptable renal function:

    a. Serum creatinine ≤1.5xULN
12. Acceptable hematologic status (without hematologic support):

    1. ANC ≥1000 cells/uL
    2. Platelet count ≥100,000/uL
    3. Hemoglobin ≥9.0 g/dL
13. All women of childbearing potential must have a negative serum pregnancy test and male and female subjects must agree to use effective means of contraception (for example, surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose.

Exclusion Criteria:

1. The subject has evidence of acute intracranial or intratumoral hemorrhage either by magnetic resonance imaging (MRI) or computerized tomography (CT) scan. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin are eligible.
2. The subject is unable or contraindicated to undergo MRI scan (e.g., has pacemaker or medically unstable).
3. The subject has not recovered to CTCAE v4.0 Grade ≤1 from AEs (except alopecia, anemia, and lymphopenia) due to antineoplastic agents, investigational drugs, or other medications that were administered prior to study.
4. The subject is pregnant or breast-feeding.
5. The subject has serious intercurrent illness, as determined by the treating physician, which would compromise either patient safety or study outcomes such as:

   * hypertension (two or more blood pressure readings performed at screening of >150 mmHg systolic or >100 mmHg diastolic) despite optimal treatment
   * active medically significant infection unresponsive to antibiotics (e.g., non- healing wound, ulcer), uncontrolled systemic infection, or bone fracture
   * clinically significant cardiac arrhythmias not controlled by appropriate medications
   * untreated hypothyroidism
   * symptomatic congestive heart failure or unstable angina pectoris within 3 months prior to study drug
   * myocardial infarction, stroke, or transient ischemic attack within 6 months prior to study drug
   * known active malignancy (other than glioma) except non-melanoma skin cancer or carcinoma in-situ in the cervix unless PI determines it would not impact patient safety or efficacy determinations
6. The subject has inherited bleeding diathesis or coagulopathy with the risk of bleeding.
7. The subject has received any of the following prior anticancer therapy:

   * Prior treatment with Bevacizumab
   * Non-standard radiation therapy such as brachytherapy, systemic radioisotope therapy, or intra-operative radiotherapy (IORT) to the target site
   * Radiation therapy within 12 weeks of screening
   * Systemic therapy (including investigational agents and small-molecule kinase inhibitors) or non-cytotoxic hormonal therapy (e.g., tamoxifen) within 14 days or 5 half-lives, whichever is shorter, prior to study start (dosing)
   * Biologic agents (antibodies, immune modulators, vaccines, cytokines) within 21 days prior to study start (dosing)
   * Nitrosoureas or mitomycin C within 42 days, or metronomic/protracted low- dose chemotherapy within 14 days, or other cytotoxic chemotherapy within 28 days, prior to study start (dosing)
   * Prior treatment with carmustine wafers
   * Patients who are currently receiving any other investigational agents and/or who have received an investigational agent in 28 days prior to study start (dosing)
8. Multifocal progression or involvement of the leptomeninges.
9. Psychiatric illness/social situations that would limit compliance with the study requirements
10. Infratentorial disease
11. The subject has a tumor located within 1-2 cm of a ventricle AND it is determined by the surgeon, PI, and sponsor to be a risk for drug extravasation to the subarachnoid space if given catheter placement and drug administration.
12. Phase 2 only: The subject should have a tumor volume of ≤20 cm3 to be included in the Phase 2 portion of the study. Subjects with tumor volumes of greater than 20 cm3 are excluded from the Phase 2 portion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2015-06-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose | 90 days
  Evaluation of any toxicity associated with research treatment per Common Toxicity Criteria for Adverse Events.
Phase 2: Overall Survival | 12 Months
  To assess overall survival (OS) following 186RNL administration by convection enhanced delivery (CED) in patients with recurrent glioma.

SECONDARY OUTCOMES:
Phase 1: Dose Distribution | Up to 7 days
  SPECT imaging of the radioactive materials spread across the tumor and surrounding brain
Phase 1: Response rate | 8 weeks followed by standard of care
  Evaluation of overall response rate by RANO criteria
Phase 1: Survival | 6 months
  Disease specific progression free survival
Phase 1: Safety of single dose of treatment | Up to 3 years
  Evaluation of any toxicity associated with research treatment as determined by the most recent version of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
Phase 2: Safety and tolerability of 186RNL | Up to 3 years
  To assess the safety and tolerability of 186RNL by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 criteria. Safety and tolerability will be defined by the percent of participants experiencing ≥ Grade 3 AE/SAE.
Phase 2: Objective response rate (ORR) | Up to 3 years.
  To determine the objective response rate (ORR) from the date of complete or partial response or Serious Treatment-Emergent Adverse Events (Safety and Tolerability)
Phase 2: Progression free survival at 6 months (PFS-6) | Up to 6 months
  To determine progression free survival at 6 months (PFS-6) as measured from the initiation of study treatment until the date of first documented progression by modified RANO criteria (recognizing the potential of pseudo progression significantly complicating the use of the RANO criteria) or date of death from any cause.
Phase 2: Progression free survival (PFS) from the initiation of study to first documented progression | Up to 3 years.
  To determine progression free survival (PFS) as measured from the initiation of study treatment until the date of first documented progression by modified RANO criteria (recognizing the potential of pseudo progression significantly complicating the use of the RANO criteria) where progression is defined as >25% in the sum of products of the perpendicular diameters of CE lesions, evidence of new lesion(s), or date of death from any cause, whichever comes first.
Phase 2: Quality of Life | Up to 3 years
  Evaluate assessing quality of life using a Quality-of-Life Questionnaire (developed in collaboration with FDA, Investigators and established glioblastoma patient advocacy groups)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Brenner, PhD, Principal Investigator — The Cancer Therapy and Research Center at UTHSCSA
Locations (3):
- United States (3):
  - Northshore University Hospital, Manhasset, New York
  - UT Southwestern Medical Center, Dallas, Texas
  - The Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas

REFERENCES:
- [Derived] Wu C, Hormuth DA 2nd, Christenson CD, Woodall RT, Abdelmalik MRA, Phillips WT, Hughes TJR, Brenner AJ, Yankeelov TE. Image-guided patient-specific optimization of catheter placement for convection-enhanced nanoparticle delivery in recurrent glioblastoma. Comput Biol Med. 2024 Sep;179:108889. doi: 10.1016/j.compbiomed.2024.108889. Epub 2024 Jul 19. PMID 39032243